CLINICAL TRIAL: NCT04970511
Title: Comparison of the Effects of Face-to-Face and Internet-Based Basic Body Awareness Therapy in Fibromyalgia Syndrome
Brief Title: Comparison of the Effects of Face-to-Face and Internet-Based BBAT in Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Özge Tahran, MSc.,Physiotherapist, Lecturer, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBAT
Record Dates: First submitted 2021-06-28; First posted 2021-07-21 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The group I: BBAT Face-to-Face Training group (Experimental): Exercises consist of supine, sitting, standing position awareness exercises and walking exercises.
  Considering eight weeks, the training is designed to progress gradually each week.
  Interventions: Behavioral: BBAT (Basic Body Awareness Therapy)
- The group II: Online BBAT training group (Experimental): Patients in the Internet-based BBAT group will conduct their training with a physiotherapist to be connected via an online video conference system.
  This group will be given the same training as the face-to-face BBAT group.
  Interventions: Behavioral: Online BBAT training
- The group III: Control group (No Intervention): No training will be applied to the control group patients.

INTERVENTIONS:
Behavioral: BBAT (Basic Body Awareness Therapy) — The group I: BBAT Face-to-Face Training (60 min) will be provided.
  Arms: The group I: BBAT Face-to-Face Training group
Behavioral: Online BBAT training — The group II: Online BBAT training (60 min) will be provided.
  Arms: The group II: Online BBAT training group

SUMMARY:
The aim of our study is to compare the effects of face-to-face and internet-based BBAT in patients diagnosed with Fibromyalgia Syndrome.

H0: Face-to-face and internet-based BBAT have superiority over each other in patients diagnosed with Fibromyalgia Syndrome.

H1: In patients diagnosed with Fibromyalgia Syndrome, face-to-face and internet-based BBAT have no superiority over each other.

DETAILED DESCRIPTION:
The aim of our study is to compare the effects of face-to-face and internet-based BBAT in patients diagnosed with Fibromyalgia Syndrome.

H0: Face-to-face and internet-based BBAT have superiority over each other in patients diagnosed with Fibromyalgia Syndrome.

H1: In patients diagnosed with Fibromyalgia Syndrome, face-to-face and internet-based BBAT have no superiority over each other.

Goals:

1. Investigation of the effects of face-to-face and internet-based BBAT on functional disability, pressure pain threshold, body awareness, posture, pain intensity, trunk position sense, postural control, balance, sleep quality, quality of life and inflammation level in patients diagnosed with Fibromyalgia Syndrome.
2. Comparison of the effects of face-to-face and internet-based BBAT on functional disability, pressure pain threshold, body awareness, posture, pain intensity, trunk position sense, postural control, balance, sleep quality, quality of life and inflammation level in patients diagnosed with Fibromyalgia Syndrome

ELIGIBILITY:
Inclusion Criteria:

1. To be between the ages of 18-65
2. Being diagnosed with FMS according to ACR 2016 criteria
3. To be diagnosed with FMS at least 6 months before the study
4. Reported pain intensity > 4 (Visual Analog Scale 0-10),
5. Individuals that do not have barriers to basic body awareness therapy.

Exclusion Criteria:

1. Pregnancy or intention to become pregnant within the study period.
2. Substance and alcohol abuse, major psychiatric disorder (preventing compliance), uncontrolled hypertension, diabetes, congestive heart failure, or other serious chronic medical condition that puts the patient at risk for the clinician to expose the patient to potentially serious consequences of their illness
3. Those who have malignancy and those receiving chemotherapy and radiotherapy causing malignancy
4. Those who have suffered from any musculoskeletal, neurological, rheumatological disorder or any condition that may interfere with evaluations (advanced respiratory or orthopedic problems such as fractures, sprains or strains, or spinal surgery) in the past 12 months -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
The Revised Fibromyalgia Impact Questionnaire (FIQR) | 8 weeks
  Limitations and functional disability in patients with fibromyalgia will be evaluated.

SECONDARY OUTCOMES:
Algometer | 8 weeks
  Pressure pain threshold measurement of characteristic 18 tender points of fibromyalgia syndrome will be performed.
Posture Screen Mobile (PSM) | 8 weeks
  Posture will be evaluated with Posture Screen Mobile (PSM), an iPad application.
The short-form McGill Pain Questionnaire | 8 weeks
  Pain will be evaluated with the short-form McGill Pain Questionnaire
Trunk repositioning error | 8 weeks
  The trunk position sense indicated by trunk reposition errors will be evaluated with the inclinometer device.
Awareness-Body-Chart=ABC | 8 weeks
  Awareness-Body-Chart=ABC will be used to assess body awareness.
Postural stability | 8 weeks
  Postural stability will be evaluated with a portable force platform.
Single Leg Balance | 8 weeks
  Balance will be evaluated with the single leg balance test with eyes open and closed.
Pittsburgh Sleep Quality Index | 8 weeks
  Sleep quality will be assessed by the Pittsburgh Sleep Quality Index.
SF-36 (the MOS 36-item short-form health survey) | 8 weeks
  As the general quality of life, the SF-36 (the MOS 36-item short-form health survey) form will be used.
Plasma Fibrinogen and Haptoglobin Protein Levels | 8 weeks
  Two plasma proteins, fibrinogen and haptoglobin, will be evaluated as markers of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Özge TAHRAN, MSc, Principal Investigator — Beykent University
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No